CLINICAL TRIAL: NCT06325995
Title: Safety and Efficacy Study of Hypofractionated Post-prostatectomy Radiotherapy (HYPORT)for Localized Prostate Cancer: a Randomized Controlled Clinical Trial
Brief Title: Hypofractionated Post-prostatectomy Radiotherapy (HYPORT)for Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Changhai HHHospital
Record Dates: First submitted 2024-03-02; First posted 2024-03-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Localized Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (COPORT) (Active Comparator): COPORT over 7 weeks.
  Interventions: Radiation: Conventional radiation therapy
- B（HYPORT） (Experimental): HYPORT over 5 weeks.
  Interventions: Radiation: Hypofractionated radiation therapy

INTERVENTIONS:
Radiation: Conventional radiation therapy — 66-74 Gy in 33-37 daily fractions of 2 Gy to the prostate bed in the absence of disease progression or unacceptable toxicity.
  Arms: A (COPORT)
Radiation: Hypofractionated radiation therapy — 57.5-65 Gy in 23-26 daily fractions of 2.5 Gy to the prostate bed in the absence of disease progression or unacceptable toxicity.
  Arms: B（HYPORT）

SUMMARY:
The aim of this trial is to compare the safety outcomes of Hypofractionated postprostatectomy radiotherapy (HYPORT) and Conventionally fractionated postprostatectomy radiotherapy(COPORT) in treating patients with localized prostate cancer.

Accumulating evidence has proven the safety and feasibility of HYPORT for localized prostate cancer.But for localized prostate cancer,the optimal dose per fraction of HYPORT is still on its way.

It is not yet known whether giving HYPORT(57.5-65 Gy in 23-26 daily fractions of 2.5 Gy ) with or COPORT may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
The present study will be conducted as a prospective, open-label, two arms clinical trial.

Patients with pathologically confirmed prostate cancer and completed radical resection of prostate cancer, will be randomized in a 1:1 ratio between arm A (COPORT) and arm B (HYPORT).

The patients in arm A will receive COPORT(66-74 Gy in 33-37 daily fractions of 2 Gy ). The patients in arm B will receive HYPORT(57.5-65 Gy in 23-26 daily fractions of 2.5 Gy ). After completion of study treatment, patients were followed up once a month for the first 3 months and once every 3 months after 3 months for a total of 5 years.

The primary endpoints of the study are toxicities parameters.The secondary endpoints include ,progression-free survival (PFS),medical economics,quality of life (QoL), overall survival (OS)and prostate cancer-specific survival period. The progression-free survival (PFS) including biochemical progression-free survival (bPFS), and radiological progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* European Cooperative Oncology Group score(ECOG):≤ 2;
* Patients with pathologically confirmed prostate cancer and completed radical resection of prostate cancer;
* Postoperative pathological staging of AJCC version 8 pT 3a, pT 3b, pT 4, margin (+), or N1; or serum PSA≥0.1 ng/ml 6 weeks after surgery; or serum PSA <0.1 ng/ml 6 weeks after surgery, subsequent follow-up process revealed two consecutive sustained PSA increases (≥0.1 ng / ml) and no clinical imaging (Whole Body Scan (ECT), magnetic resonance imaging (MRI),68Ga PSMA PET / CT, etc.) signs of metastasis;
* Expected survival time >5 years;
* Patients who voluntarily accept the experimental study protocol after informing the existing treatment options;

Exclusion Criteria:

* poor recovery of postoperative urinary control;
* a previous history of pelvic and abdominal radiotherapy;
* Participate in other clinical trials that are mutually exclusive with the study intervention within 4 weeks prior to the start of the study;
* Patients with other malignancies and acute or chronic infections such as human immunodeficiency virus (HIV) (+), hepatitis C virus (HCV) (+) and/or positive syphilis;
* Patients that the investigator considers unsuitable to participate in the clinical trial; patients with other serious systemic diseases, evaluation and compliance of the trial, including severe respiratory, circulatory, neurological, mental, digestive, endocrine, immune, urinary, and other systemic diseases;
* Patients with contraindications related to radiotherapy;
* Written informed consent could not be provided, and treatment compliance was poor.Patients unsuitable for participation in this clinical trial as per the judgement of the investigator.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiotherapy-related gastrointestinal and urogenital tract adverse events | Assessment toxicities parameters at 5 years
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0

SECONDARY OUTCOMES:
5-year progression-free survival (PFS) | Assessment progression-free survival (PFS) at 5 years
  To assess progression-free survival (PFS) including biochemical progression-free survival (bPFS), and radiological progression-free survival.
quality of life (QoL) | through study completion, an average of 5 years
  Expanded Prostate Cancer Index (EPIC-26)：The EPIC is a prostate cancer health-related quality of life (HRQOL) self-administered instrument measuring patient-reported urinary, bowel, sexual, and hormonal symptoms related to prostate cancer treatments. Response options for each item form a Likert scale with scores transformed linearly to a 0-100 scale. Domain scores are also on a 0-100 scale with higher scores representing better HRQOL.
medical expenses | Assessment the medical economics during the treatment,up to 7 weeks
  The medical expenses during the time of interventions.The medical expenses include the payments of doctor and hospital visits, co-pays, radiotherapy and so on.
Overall survival (OS) | Assessment overall survival (OS) at 5 years
  To assess the overall survival (OS)
Prostate cancer-specific survival | Assessment prostate cancer-specific survival at 5 years
  To assess the prostate cancer-specific survival
Physical Activity Rank Scale-3 (ARS-3) | through study completion, an average of 5 years
  To assess the physical activity rank.The scale was compiled by Japanese psychologist KIMIO HASHIMOTO and introduced and revised by Liang Deqing from Wuhan Physical Education University. There are only 3 items in this scale, which adopts 5 grades from 1 to 5, and examines the level of physical activity from 3 aspects: intensity, time and frequency of participating in physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics,treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol
Time Frame: Within 5 years after the publication of the study.
Access Criteria: Data may be shared with radiation oncologists and specialists in surgery who are interested in examining the efficacy and toxicity of localized prostate cancer treated with HYPORT or COPORT. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.